CLINICAL TRIAL: NCT03002298
Title: Motor Learning From Virtual to Natural Environments in Individuals With Duchenne Muscular Dystrophy
Brief Title: Virtual Reality in Individuals With Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16796513.1.0000.0065
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DMD gesture task (Experimental): Experimental group that made the task using a gesture in front of a webcam
  Interventions: Behavioral: DMD gesture task
- DMD button-press task (Experimental): Experimental group that made the task pressing the button
  Interventions: Behavioral: DMD button-press task
- Control group gesture task (Active Comparator): Control group that made the task using a gesture in front of a webcam
  Interventions: Behavioral: Control group gesture task
- Control group button-press task (Active Comparator): Control group that made the task pressing the button
  Interventions: Behavioral: Control group button-press task

INTERVENTIONS:
Behavioral: DMD gesture task — Timing coincident task in a virtual environment, using motor learning protocol in which a gesture in front of a webcam shoub be done to reach the task
  Arms: DMD gesture task
Behavioral: DMD button-press task — Timing coincident task in a virtual environment, using motor learning protocol in which the task shoub be done by pressing a button on the keyboard
  Arms: DMD button-press task
Behavioral: Control group gesture task — Timing coincident task in a virtual environment, using motor learning protocol in which a gesture in front of a webcam shoub be done to reach the task
  Arms: Control group gesture task
Behavioral: Control group button-press task — Timing coincident task in a virtual environment, using motor learning protocol in which the task shoub be done by pressing a button on the keyboard
  Arms: Control group button-press task

SUMMARY:
With the growing accessibility of computer-assisted technology, one option for rehabilitation programs for individuals with Duchenne muscular dystrophy (DMD) is the use of virtual reality environments to enhance motor practice. Thus, it is important to examine whether performance improvements in the virtual environment generalize to the natural environment. To examine this issue, we had 64 individuals, 32 of which were individuals with DMD and 32 were typically developing individuals. The groups practiced two coincidence timing tasks. In the more tangible button-press task, the individuals were required to 'intercept' a falling virtual object at the moment it reached the interception point by pressing a key on the computer. In the more abstract task, they were instructed to 'intercept' the virtual object by making a hand movement in a virtual environment using a webcam.

DETAILED DESCRIPTION:
The Department of Electronic System Engineering of the Polytechnic School of the University of São Paulo (Brazil) developed the software that superimposes virtual objects over images of real world, captured with a webcam.

The coincidence timing task could either have a virtual or a real interface. For the real interface, a keyboard was used. For the virtual interface, a webcam recorded a marker on the table alongside the keyboard of the computer. The images were fed into the computer and analyzed online. Using the custom-made software, it was determined whether or not the participant's hand occluded the marker, which was then fed back to the virtual environment. The coincidence timing task was based on the Bassin Anticipation Timer. To this end, 10 3D-cubes were displayed simultaneously in a vertical column on a monitor. The cubes were turned on (i.e., they changed from white to green) and off sequentially (from top to bottom) until the target cube (i.e., the tenth cube) was reached. The task for the participant was to either press the space bar on the keyboard (i.e., tangible button press task, by physical contact, represented on figure 1A and 1B) or to make a sideward hand gesture as if hitting the target object (i.e., the more abstract gesture task, with no physical contact, represented on the figure 1C and 1D), i.e., occluding the marker at the exact moment the target cube turned green.

Participants performed the task individually in a quiet room with only the examiner who gave the instructions present. The computer was placed on a table. The participants were seated in their wheelchair, which was adjusted according to the needs of the individual.

The examiner explained the task verbally and gave three demonstrations of how to perform the coincidence timing tasks. The participants were instructed to place the preferred hand (i.e., the less affected hand) on a mark aside to the target (The location was individually adjusted but ranged from 2 to 4 cm from the target). Once the first top cube turned on, the individual had to move his hand to either touch the target key on the keyboard or to make a hitting gesture in front of the webcam, exactly at the moment coinciding with the bottom target cube turning on. Different sounds were provided as feedback for either a hit or miss during acquisition, retention and transfer, the range of error being -200 to 200ms.

Participants with DMD and TD were divided into two subgroups randomly: (a) button-press task group (BPT) - in this group during the acquisition phase the participants should press the space button on keyboard to complete the coincidence timing task (more real interface) and (b) gesture task group (GT) - in this group during the acquisition phase the participants should cross a virtual target created by a webcam to complete the coincidence timing task instead of press the computer button (more virtual interface).

For all tasks (button-press and gesture), during the acquisition phase, all groups started performing 20 attempts of the coincidence timing task and, after five minutes with no contact with the task, they performed five more repetitions for the retention phase (both phases in slower speed - with the turning on and off of the lights in an interval of 400ms), finally they performed five repetitions for two different transfers phases: the first transfer was performed with a faster speed - 300ms of lights interval (transfer with speed increase - TSI). The second transfer was performed with change task (transfer with exchange of en vironment - TEE) between groups by doing 5 attempts transfer phase in another interface. It means, the group that has done the acquisition phase in button-press task performed the transfer on gesture task and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of Duchenne Muscular Dystrophy confirmed by molecular method and/or protein expression in skeletal muscle;
* signing of an informed consent form from the individual or person legally responsible.

Exclusion Criteria:

* presence of associated comorbidities;
* inability in comprehension of the task.

Ages: 12 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Motor Learning test by using a timing coincident task in virtual reality | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: Undecided